CLINICAL TRIAL: NCT06553755
Title: Unraveling the Multidimensional Functional Recovery Patterns and Prognostic Factors in Post-Discharged Stroke Survivors: A Retrospective Study
Brief Title: Multidimensional Recovery Patterns and Prognostic Factors After Stroke
Status: Active, not recruiting | Type: Observational
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Feng-Hang Chang, Professor, Taipei Medical University
Other Study IDs: N202406014
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: functional status; prognosis; recovery; social participation; stroke subtypes
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to compare the 1-year recovery trajectories of multidimensional functional recovery among stroke survivors after discharge from hospital care.

To address this purpose, a retrospective analysis will be conducted using clinical data from two independent cohorts derived from previously published prospective observational studies. The study will conduct generalized estimating equations and mixed-effects regression models to assess differences in recovery trends among stroke subgroups.

The findings will provide detailed profiles of longitudinal changes in functional outcomes one year after discharge from hospital care. These results will clarify how stroke subtypes influence long-term functional outcomes and will guide the development of targeted interventions.

DETAILED DESCRIPTION:
Different stroke types have unique pathophysiological mechanisms that likely affect various recovery outcomes. Understanding stroke-subtype-specific functional recovery and outcomes is crucial for effective rehabilitation and discharge planning. However, current evidence does not fully reveal how functional outcomes differ by stroke subtype, leaving gaps in our understanding of how these differences impact post-stroke recovery. Identifying the specific recovery patterns and prognostic factors associated with each stroke subtype can enhance personalized rehabilitation strategies and improve patient care.

To address this purpose, a retrospective study utilizing clinical data from two independent cohorts recruited from collaborative hospitals in Northern Taiwan between 2016 and 2018 will be implemented. The study will employ several outcome measures, including the Participation Measure-3 Domains, 4 Dimensions (PM-3D4D), the Activity Measure for Post-Acute Care (AM-PAC), the modified Rankin Scale (mRS) and other standardized assessment tools. Participants will be assessed from hospital discharge until 12-month follow-up. Data analysis will use generalized estimating equations and mixed-effects regression models to evaluate differences in recovery trends among stroke subgroups.

The findings will offer comprehensive insights into the progression of various functional outcomes of specific stroke subtypes over the course of one year following discharge. The study will also identify factors associated with long-term functional outcomes and investigate how those factors impact the trend of functional recovery. These results will demonstrate the association of stroke subtypes and long-term functional outcomes, facilitating the development of targeted interventions.

ELIGIBILITY:
Inclusion Criteria:

Stroke survivors

1. aged 20 years or older;
2. were diagnosed with a stroke confirmed by physicians;
3. were assessed at least one of the outcomes of interest, including participation (Participation Measure-3 Domains, 4 Dimensions, PM-3D4D), activity limitations (Activity Measure for Post-Acute Care short forms, AM-PAC), HRQoL (EuroQol-5D-3L, EQ-5D-3L), and cognitive impairments (Montreal Cognitive Assessment, MoCA).

Exclusion Criteria: Stroke survivors who missed all follow-up assessments.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The retrospective study is based on the clinical data of two independent cohorts from previously published prospective, observational studies. The ethics committee approved these studies at the Taipei Medical University. Both cohorts recruited stroke patients at three hospitals (Taipei Medical University Hospital, Wan Fang Hospital, Shuang Ho Hospital) between January 2016 and September 2018, collecting functional outcomes and person-environment variables since discharged from hospital to 12-month post-discharge follow-up.
Sampling Method: Probability Sample
Enrollment: 1270 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Participation Measure-3 Domains, 4 Dimensions (PM-3D4D) | From discharged from acute care up to 1 year
  The PM-3D4D is a 24-item measure that was designed to evaluate three domains of participation: Productivity, Social, and Community. Respondents are asked to rate each item on four dimensions: (1) 'Diversity of participation' (yes [1] vs. no [0]); (2) 'Frequency'(5- and 7-point scales, from "never" to "everyday or almost everyday"); (3) 'Desire for change' (yes [1] vs. no[0]); and (4) 'Perceived difficulty' (4-point scale, from "very difficult" [1] to "not difficult at all" [4]). Each dimensional score of the PM-3D4D can be separately summed for each domain. Psychometric properties of the PM-3D4D were established in rehabilitation populations.
Activity Measure for Post-Acute Care (AM-PAC) | From discharged from acute care up to 1 year
  The Activity Measure for Post-Acute Care (AMPAC) Outpatient Short Forms consists of three subscales that assesses three activity domains: basic mobility (18 items), daily activity (15 items), and applied cognitive (19 items). Each item asks the respondent to rate the difficulty to perform specified activities using a 4-point scale. The summary scores range 18-72, 15-60, 19-76 points respectively among three subscales. Higher score indicates better function of the specific domain. The summary scores for each subscale will be transformed into standardized scores on the t-score scale.
Euro-QoL-5-Dimension-3 Level (EQ-5D-3L) | From discharged from acute care up to 1 year
  The Euro-QoL-5-Dimension-3 Level (EQ-5D-3L) is used to assess participant's health related quality of life which consist of 5 ordinal scale items and 1 item with visual analog scale. Ordinal scales are rated 0-3 points with higher score indicating the pooer health-related quality of life. visual analog scale are rated by respondents reporting perceived health status with a grade ranging from 0 to 100 with higher score indicating the better health status).
Montreal Cognitive Assessment (MoCA) | From discharged from acute care up to 1 year
  Montreal Cognitive Assessment (MoCA) is a clinician-reported measure consisting of cognition domains such as: visuospatial skills, executive functions, attention, concentration, calculation, language, abstraction, memory, and orientation. The summary score ranges from 0-30 points with higher scores indicating better cognitive function.

SECONDARY OUTCOMES:
Barthel Index (BI) | From discharged from acute care up to 1 year
  Barthel Index (BI) is a commonly used measurement indicating independence level of self-care, with higher scores indicating a better self-care independence.
Modified Rankin Scale (mRS) | From discharged from acute care up to 1 year
  The modified Rankin Scale (mRS) is designed to measure functional status after a stroke. Each participant is rated 0-6 point on an ordinal scale with lower score indicating greater functional status after stroke.
The Center for Epidemiologic Studies Depression Scale (CES-D) | From discharged from acute care up to 1 year
  The Center for Epidemiologic Studies Depression Scale (CES-D) is a self-reported outcome measure of depressive symptoms, with higher scores indicating the presence of more severe symptom (range: 0-60).

OTHER OUTCOMES:
National Institutes of Health Stroke scale (NIHSS) | From discharged from acute care up to 1 year
  National Institutes of Health Stroke scale (NIHSS) is a 15-item measurement designed to assess neurological symptoms
Personal factors | From discharged from acute care up to 1 year
  General information relating to stroke individuals, including age of onset, sex, diagnosis, time since onset, comobidities, education, marital status, monthly income, etc.
Environmental factors | From discharged from acute care up to 1 year
  Information relating to the environments in which the stroke individuals live, including living with caregiver(s), house with/without a elevator, social support, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan